CLINICAL TRIAL: NCT02301156
Title: A Phase 3, Randomized, Study to Assess the Efficacy and Safety of Ublituximab in Combination With Ibrutinib Compared to Ibrutinib Alone, in Patients With Previously Treated High-Risk Chronic Lymphocytic Leukemia (CLL)
Brief Title: Ublituximab in Combination With Ibrutinib Versus Ibrutinib Alone in Participants With Previously Treated High-Risk Chronic Lymphocytic Leukemia (CLL)
Acronym: GENUINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UTX-IB-301
Record Dates: First submitted 2014-11-20; First posted 2014-11-25 (Estimated); Results first posted 2022-05-20 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-04

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ublituximab; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Ublituximab + Ibrutinib (Experimental): Participants will receive ublituximab intravenous (IV) infusion, up to 150 milligrams (mg) once on Day 1, 750 mg on Day 2, 900 mg on Days 8 and 15 of Cycle 1 (Cycle duration=28 days) followed by 900 mg on Day 1 of Cycles 2 to 6 and 900 mg on Day 1 of every 3rd cycle thereafter for up to 62 months along with ibrutinib 420 mg capsules, orally, once daily (QD) in each 28-day cycle for up to 62 months.
  Interventions: Drug: Ublituximab; Drug: Ibrutinib
- Ibrutinib (Active Comparator): Participants will receive ibrutinib 420 mg capsules, orally, QD in each 28-day cycle up to 62 months.
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ublituximab — Administered as an IV infusion
  Other Names: TG-1101
  Arms: Ublituximab + Ibrutinib
Drug: Ibrutinib — Administered orally
  Other Names: IMBRUVICA

SUMMARY:
This study evaluates the effect of the addition of ublituximab, a novel monoclonal antibody, to ibrutinib compared to ibrutinib alone on antitumor activity, as measured by the overall response rate (ORR = CR [complete response] + PR [partial response]) in previously treated Chronic Lymphocytic Leukemia (CLL) participants with high-risk cytogenetic features. Half of the participants will receive ublituximab in combination with ibrutinib, while the other half will receive ibrutinib alone.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated Chronic Lymphocytic Leukemia (CLL) requiring treatment
* At least one high-risk cytogenetic feature defined by the presence of 17p deletion, 11q deletion and/or p53 mutation
* Eastern Cooperative Oncology Group (ECOG) score of 0 to 2

Exclusion Criteria:

* Any major surgery, chemotherapy or immunotherapy within the last 21 days
* Evidence of hepatitis B virus, hepatitis C virus or known human immunodeficiency virus (HIV) infection
* Autologous hematologic stem cell transplant within 3 months of study entry. Prior Allogeneic hematologic stem cell transplant is excluded
* Transformation of CLL to aggressive Non-Hodgkin's Lymphoma (NHL) (Richter's transformation)
* Previous therapy with ibrutinib, or any drug that specifically inhibits Bruton's tyrosine kinase (BTK)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2015-01-27 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Sharman, MD, Study Chair — Willamette Valley Cancer Institute
Locations (85):
- United States (84):
  - TG Therapeutics Investigational Trial Site, Huntsville, Alabama
  - TG Therapeutics Investigational Trial Site, Mobile, Alabama
  - TG Therapeutics Investigational Trial Site, Chandler, Arizona
  - TG Therapeutics Investigational Trial Site, Tucson, Arizona
  - TG Therapeutics Investigational Trial Site, Fayetteville, Arkansas
  - TG Therapeutics Investigational Trial Site, Jonesboro, Arkansas
  - TG Therapeutics Investigational Trial Site, Fullerton, California
  - TG Therapeutics Investigational Trial Site, Greenbrae, California
  - TG Therapeutics Investigational Trial Site, Los Angeles, California
  - TG Therapeutics Investigational Trial Site, Pismo Beach, California
  - TG Therapeutics Investigational Trial Site, Pleasanton, California
  - TG Therapeutics Investigational Trial Site, Santa Barbara, California
  - TG Therapeutics Investigational Trial Site, Aurora, Colorado
  - TG Therapeutics Investigational Trial Site, Bridgeport, Connecticut
  - TG Therapeutics Investigational Trial Site, Stamford, Connecticut
  - TG Therapeutics Investigational Trial Site, Newark, Delaware
  - TG Therapeutics Investigational Trial Site, Boca Raton, Florida
  - TG Therapeutics Investigational Trial Site, Fort Myers, Florida
  - TG Therapeutics Investigational Trial Site, Orange City, Florida
  - TG Therapeutics Investigational Trial Site, Pensacola, Florida
  - TG Therapeutics Investigational Trial Site, St. Petersburg, Florida
  - TG Therapeutics Investigational Trial Site, West Palm Beach, Florida
  - TG Therapeutics Investigational Trial Site, Albany, Georgia
  - TG Therapeutics Investigational Trial Site, Newnan, Georgia
  - TG Therapeutics Investigational Trial Site, Evanston, Illinois
  - TG Therapeutics Investigational Trial Site, Maywood, Illinois
  - TG Therapeutics Investigational Trial Site, Niles, Illinois
  - TG Therapeutics Investigational Trial Site, Urbana, Illinois
  - TG Therapeutics Investigational Trial Site, Fort Wayne, Indiana
  - TG Therapeutics Investigational Trial Site, Indianapolis, Indiana
  - TG Therapeutics Investigational Trial Site, Ames, Iowa
  - TG Therapeutics Investigational Trial Site, Cedar Rapids, Iowa
  - TG Therapeutics Investigational Trial Site, Westwood, Kansas
  - TG Therapeutics Investigational Trial Site, Baton Rouge, Louisiana
  - TG Therapeutics Investigational Trial Site, New Orleans, Louisiana
  - TG Therapeutics Investigational Trial Site, Baltimore, Maryland
  - TG Therapeutics Investigational Trial Site, Bethesda, Maryland
  - TG Therapeutics Investigational Trial Site, Columbia, Maryland
  - TG Therapeutics Investigational Trial Site, Salisbury, Maryland
  - TG Therapeutics Investigational Trial Site, Boston, Massachusetts
  - TG Therapeutics Investigational Trial Site, Springfield, Massachusetts
  - TG Therapeutics Investigational Trial Site, Worcester, Massachusetts
  - TG Therapeutics Investigational Trial Site, Detroit, Michigan
  - TG Therapeutics Investigational Trial Site, Coon Rapids, Minnesota
  - TG Therapeutics Investigational Trial Site, Saint Louis Park, Minnesota
  - TG Therapeutics Investigational Trial Site, Lincoln, Nebraska
  - TG Therapeutics Investigational Trial Site, Omaha, Nebraska
  - TG Therapeutics Investigational Trial Site, Lebanon, New Hampshire
  - TG Therapeutics Investigational Trial Site, East Brunswick, New Jersey
  - TG Therapeutics Investigational Trial Site, Howell Township, New Jersey
  - TG Therapeutics Investigational Trial Site, Morristown, New Jersey
  - TG Therapeutics Investigational Trial Site, Pompton Plains, New Jersey
  - TG Therapeutics Investigational Trial Site, Somerville, New Jersey
  - TG Therapeutics Investigational Trial Site, New York, New York
  - TG Therapeutics Investigational Trial Site, Syracuse, New York
  - TG Therapeutics Investigational Trial Site, Charlotte, North Carolina
  - TG Therapeutics Investigational Trial Site, Durham, North Carolina
  - TG Therapeutics Investigational Trial Site, Raleigh, North Carolina
  - TG Therapeutics Investigational Trial Site, Canton, Ohio
  - TG Therapeutics Investigational Trial Site, Cincinnati, Ohio
  - TG Therapeutics Investigational Trial Site, Cleveland, Ohio
  - TG Therapeutics Investigational Trial Site, Portland, Oregon
  - TG Therapeutics Investigational Trial Site, Springfield, Oregon
  - TG Therapeutics Investigational Trial Site, Camp Hill, Pennsylvania
  - TG Therapeutics Investigational Trial Site, Philadelphia, Pennsylvania
  - TG Therapeutics Investigational Trial Site, Pawtucket, Rhode Island
  - TG Therapeutics Investigational Trial Site, Greenville, South Carolina
  - TG Therapeutics Investigational Trial Site, Sioux Falls, South Dakota
  - TG Therapeutics Investigational Trial Site, Watertown, South Dakota
  - TG Therapeutics Investigational Trial Site, Memphis, Tennessee
  - TG Therapeutics Investigational Trial Site, Nashville, Tennessee
  - TG Therapeutics Investigational Trial Site, Austin, Texas
  - TG Therapeutics Investigational Trial Site, Dallas, Texas
  - TG Therapeutics Investigational Trial Site, Denton, Texas
  - TG Therapeutics Investigational Trial Site, Fort Sam Houston, Texas
  - TG Therapeutics Investigational Trial Site, San Antonio, Texas
  - TG Therapeutics Investigational Trial Site, Tyler, Texas
  - TG Therapeutics Investigational Trial Site, Webster, Texas
  - TG Therapeutics Investigational Trial Site, Ogden, Utah
  - TG Therapeutics Investigational Trial Site, Blacksburg, Virginia
  - TG Therapeutics Investigational Trial Site, Richmond, Virginia
  - TG Therapeutics Investigational Trial Site, Seattle, Washington
  - TG Therapeutics Investigational Trial Site, Spokane, Washington
  - TG Therapeutics Investigational Trial Site, Vancouver, Washington
- TG Therapeutics Investigational Trial Site, Ashkelon, Israel

IPD SHARING:
Plan to Share IPD: No
TG Therapeutics does not currently plan to share IPD.

REFERENCES:
- [Derived] Sharman JP, Brander DM, Mato AR, Ghosh N, Schuster SJ, Kambhampati S, Burke JM, Lansigan F, Schreeder MT, Lunin SD, Zweibach A, Shtivelband M, Travis PM, Chandler JC, Kolibaba KS, Sportelli P, Miskin HP, Weiss MS, Flinn IW. Ublituximab plus ibrutinib versus ibrutinib alone for patients with relapsed or refractory high-risk chronic lymphocytic leukaemia (GENUINE): a phase 3, multicentre, open-label, randomised trial. Lancet Haematol. 2021 Apr;8(4):e254-e266. doi: 10.1016/S2352-3026(20)30433-6. Epub 2021 Feb 22. PMID 33631112

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 126 participants were enrolled at investigative sites in Israel and the United States (US) from 27 January 2015 to 01 April 2020.
Pre-assignment Details: Participants with previously treated Chronic Lymphocytic Leukemia (CLL) who had at least one high-risk cytogenetic abnormality were enrolled and randomized in a 1:1 ratio to receive either ublituximab in combination with ibrutinib or ibrutinib alone.
Groups:
- Ublituximab + Ibrutinib: Participants received ublituximab intravenous (IV) infusion, up to 150 milligrams (mg) once on Day 1, 750 mg on Day 2, 900 mg on Days 8 and 15 of Cycle 1 (Cycle duration=28 days) followed by 900 mg on Day 1 of Cycles 2 to 6 and 900 mg on Day 1 of every 3rd cycle thereafter for up to 54.6 months along with ibrutinib 420 mg capsules, orally, once daily (QD) in each 28-day cycle for up to 51.6 months.
- Ibrutinib: Participants received ibrutinib 420 mg capsules, orally, QD in each 28-day cycle up to 56.3 months.
Period: Overall Study
Arm/Group | Ublituximab + Ibrutinib | Ibrutinib
Started | 64 | 62
Intent to Treat (ITT) Population (Intent-to-treat (ITT) Population included all randomized participants.) | 64 | 62
Safety Population (Safety Population included all participants who received at least one dose of study medication (ublituximab + ibrutinib or ibrutinib alone).) | 59 | 58
Completed | 11 | 10
Not Completed | 53 | 52
Not completed — Adverse Event | 13 | 14
Not completed — Death | 1 | 5
Not completed — Investigator Decision (includes non-compliance with study drug, investigator determined suitability) | 2 | 2
Not completed — Site Terminated by Sponsor at the End of Study | 27 | 16
Not completed — Withdrawal of Consent by Subject | 4 | 12
Not completed — Reason not Specified | 6 | 3

BASELINE CHARACTERISTICS:
Population: ITT Population included all randomized participants.
Groups:
- Ublituximab + Ibrutinib: Participants received ublituximab IV infusion, up to 150 mg once on Day 1, 750 mg on Day 2, 900 mg on Days 8 and 15 of Cycle 1 (Cycle duration=28 days) followed by 900 mg on Day 1 of Cycles 2 to 6 and 900 mg on Day 1 of every 3rd cycle thereafter for up to 54.6 months along with ibrutinib 420 mg capsules, orally, QD in each 28-day cycle for up to 51.6 months.
- Total: Total of all reporting groups
Arm/Group | Ublituximab + Ibrutinib | Ibrutinib | Total
Number analyzed (Participants) | 64 | 62 | 126
Age, Continuous [Mean (Full Range); unit: years] | 67.0 [42 to 86] | 67.2 [51 to 85] | 67.1 [42 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 16 | 36
  Male | 44 | 46 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 62 | 59 | 121
  Unknown or Not Reported | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 6 | 13
  White | 56 | 55 | 111
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Israel | 1 | 0 | 1
  United States | 63 | 62 | 125

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR: Percentage of participants with best overall response of partial response(PR) and complete response(CR). CR criteria: No evidence of new disease; Absolute lymphocyte count(ALC)<4x10^9/liter(L); Regression of all target nodal masses to ≤1.5 centimeters(cm) in longest diameter(LD); Normal spleen,liver size; Regression to normal of all nodal non-target disease and disappearance of all detectable; Non-nodal, non-target disease; Morphologically negative bone marrow; No lymphoid nodules; Absolute neutrophil count(ANC)>1.5x10^9/L,platelets≥100x10^9/L,hemoglobin (Hgb)≥110 gram per liter(g/L). PR criteria: No evidence of new disease; Response in 2 of following if abnormal at baseline: ALC<4x10^9/L or >=50% decrease from baseline in sum of products(SPD) of target nodal lesions; splenomegaly; hepatomegaly;>=50% decrease from baseline in CLL marrow infiltrate/B-lymphoid nodules; response in any 1:ANC>1.5x10^9/L,platelets>100x10^9/L,Hgb>110g/L or >=50% increase over baseline in any of these.
Time Frame: Up to 62 months
Population: ITT Population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Ublituximab + Ibrutinib | Ibrutinib
Number analyzed (Participants) | 64 | 62
percentage of participants | 84.4 | 69.4
Statistical Analysis 1: Comparison: Ublituximab + Ibrutinib vs Ibrutinib; Test type: Superiority; p = 0.0463, Cochran-Mantel-Haenszel; P-value was estimated by Cochran-Mantel-Haenszel (CMH) test stratified by the randomization strata prior lines of therapy

2. Secondary Outcome: Complete Response (CR) Rate
Description: The CR rate was defined as the percentage of participants who achieved CR. CR criteria: No evidence of new disease; ALC <4 x 10^9/L; Regression of all target nodal masses to normal size ≤1.5 cm in the LD; Normal spleen and liver size; Regression to normal of all nodal non-target disease and disappearance of all detectable; Non-nodal, non-target disease; Morphologically negative bone marrow; No lymphoid nodules; ANC >1.5 x 10^9/L, platelets ≥100 x 10^9/L, Hgb ≥110 g/L.
Time Frame: Up to 62 months
Population: ITT Population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Ublituximab + Ibrutinib | Ibrutinib
Number analyzed (Participants) | 64 | 62
percentage of participants | 18.8 | 4.8
Statistical Analysis 1: Comparison: Ublituximab + Ibrutinib vs Ibrutinib; Test type: Superiority; p = 0.0159, Cochran-Mantel-Haenszel; P-value was estimated by CMH test stratified by the randomization strata prior lines of therapy

3. Secondary Outcome: Minimum Residual Disease (MRD) Negativity Rate
Description: MRD negativity rate was defined as the percentage of participants who were MRD negative post-baseline. If a participant was determined to be MRD negative by peripheral blood, a bone marrow aspirate was obtained to assess MRD in the bone marrow.
Time Frame: Up to 62 months
Population: ITT Population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ublituximab + Ibrutinib | Ibrutinib
Number analyzed (Participants) | 64 | 62
percentage of participants | 45.3 [32.8 to 58.3] | 9.7 [3.6 to 19.9]
Statistical Analysis 1: Comparison: Ublituximab + Ibrutinib vs Ibrutinib; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; P-value was estimated using CMH test stratified by the randomization strata prior lines of therapy; Rate Difference = 35.64, 95% CI 2-sided [21.39 to 49.88] — 95% Confidence Interval (CI) was estimated using Clopper-Pearson method based on the binomial distribution

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from the date of randomization until the date of first documentation of definitive disease progression (PD) or date of death from any cause, whichever occurs first. PD requires at least one of the following: New nodes >1.5 cm in the LD and >1.0 in longest perpendicular diameter (LPD), new or recurrent hepatomegaly or splenomegaly, new or reappearance of an unequivocal extra-nodal lesion, ≥50% increase from the nadir in the sum of products of target lesions, ≥50% increase in the LD of an individual node or extra-nodal mass, splenic/hepatic enlargement of ≥50% from nadir, unequivocal increase in the size of non-target disease, transformation to a more aggressive histology, decrease in platelet count or Hgb, >50% decrease from the highest on-study platelet count, >20 g/L decrease from the highest on-study Hgb.
Time Frame: From the randomization until the first documentation of PD or death whichever occurs first or up to 62 months
Population: ITT Population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ublituximab + Ibrutinib | Ibrutinib
Number analyzed (Participants) | 64 | 62
months | NA [NA to NA] — Median, upper and lower limit of 95% CI were not estimable due to low number of participants with event. | 47.2 [18.9 to NA] — Upper limit of 95% CI was not estimable due to low number of participants with event.
Statistical Analysis 1: Comparison: Ublituximab + Ibrutinib vs Ibrutinib; Test type: Superiority; p = 0.0961, Log Rank; P-value was estimated by stratified log rank test and the stratification was based on the randomization strata prior lines of therapy; Hazard Ratio (HR) = 0.573, 95% CI 2-sided [0.295 to 1.113] — Stratified Hazard Ratio and 95% CI were estimated using Cox proportion hazard model and the stratification was based on the randomization strata prior lines of therapy

5. Secondary Outcome: Duration of Response (DOR)
Description: DOR:Interval from first documentation of CR/PR to first documentation of PD or death from any cause.CR:ALC<4x10^9/L;Regression to normal of target nodal masses,nodal non-target disease,and no detectable non-nodal,non-target disease;Normal spleen,liver size;Morphologically negative bone marrow,No lymphoid nodules;ANC>1.5x10^9/L,Platelets≥100x10^9/L,Hgb≥110 g/L.PR:Response in 2 or more:ALC<4x10^9/L,>=50% drop from baseline in ALC or SPD of target nodal lesions,Hepatosplenomegaly,>=50% decrease from baseline in CLL marrow infiltrate/B-lymphoid nodules;Response in 1 or more:ANC>1.5x10^9/L,Platelets>100x10^9/L,Hgb>110 g/L or >=50% increase over baseline in any.PD:Response in 1 or more:new nodes,Hepatosplenomegaly,unequivocal extra-nodal lesion;≥50% increase from nadir in SPD of target lesions or LD of node/extra-nodal mass or Splenic/Hepatic size,Unequivocal increase in non-target disease,More aggressive histology;Drop of >50% in platelets/>20g/L in Hgb from highest on-study count.
Time Frame: From the first dose of study drug until the first documentation of PD or death whichever occurs first or up to 62 months
Population: Participants in the ITT Population (included all randomized participants) who achieved either CR or PR were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ublituximab + Ibrutinib | Ibrutinib
Number analyzed (Participants) | 54 | 43
months | NA [NA to NA] — Median, upper and lower limit of 95% CI were not estimable due to low number of participants with event. | 39.1 [16.7 to NA] — Upper limit of 95% CI was not estimable due to low number of participants with event.
Statistical Analysis 1: Comparison: Ublituximab + Ibrutinib vs Ibrutinib; Test type: Superiority; p = 0.1486, Log Rank; [statistical method as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.569, 95% CI 2-sided [0.263 to 1.234] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Time to Response (TTR)
Description: TTR was defined as the interval from the randomization to the first documentation of CR or PR. CR criteria: No evidence of new disease; ALC <4 x 10^9/L; Regression of all target nodal masses to normal size ≤1.5 cm in the LD; Normal spleen and liver size; Regression to normal of all nodal non-target disease and disappearance of all detectable; Non-nodal, non-target disease; Morphologically negative bone marrow; No lymphoid nodules; ANC >1.5 x 10^9/L, platelets ≥100 x 10^9/L, Hgb ≥110 g/L. PR criteria: No evidence of new disease; Response in 2 of following when abnormal at baseline: ALC<4 x 10^9/L or >=50% decrease from baseline in SPD of target nodal lesions; splenomegaly; hepatomegaly; >=50% decrease from baseline in CLL marrow infiltrate/B-lymphoid nodules; and Response in 1 of the following: ANC>1.5 x 10^9/L, platelets>100 x 10^9/L, Hgb>110 g/L or >=50% increase over baseline in any of these.
Time Frame: From the randomization up to 62 months
Population: Participants in the ITT Population (included all randomized participants) who achieved either CR or PR were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ublituximab + Ibrutinib | Ibrutinib
Number analyzed (Participants) | 54 | 43
months | 2.0 [2.0 to 2.1] | 3.9 [2.2 to 8.3]
Statistical Analysis 1: Comparison: Ublituximab + Ibrutinib vs Ibrutinib; Test type: Superiority; p = 0.0004, Log Rank; [statistical method as in outcome 4, analysis 1]; Hazard Ratio (HR) = 2.163, 95% CI 2-sided [1.399 to 3.344] — [estimate comment as in outcome 4, analysis 1]

7. Secondary Outcome: Percentage of Participants Experiencing at Least One Treatment-Emergent Adverse Event (TEAE)
Description: An adverse event (AE) is any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporarily associated with the use of a medicinal product, whether or not considered related to the medicinal product. TEAE is any AE that occur after first dosing of study medication and through the end of the study or through 30 days after the last dose of study treatment, or is considered treatment-related regardless of the start date of the event, or is present before first dosing of study medication but worsens in intensity or the investigator subsequently considers treatment-related.
Time Frame: From the first dose up to 30 days after the last dose of study drug (up to 57.3 months)
Population: Safety Population included all participants who received at least one dose of study medication (ublituximab + ibrutinib or ibrutinib alone).
Measure: Number; unit: percentage of participants
Arm/Group | Ublituximab + Ibrutinib | Ibrutinib
Number analyzed (Participants) | 59 | 58
percentage of participants | 100 | 100

ADVERSE EVENTS:
Time Frame: Adverse Events: From the first dose up to 30 days after the last dose of study drug (up to 57.3 months); All-Cause Mortality: From the first dose up to end of study (up to 62 months)
Description: Safety Population included all participants who received at least one dose of study medication (ublituximab + ibrutinib or ibrutinib alone).
Arm/Group | Ublituximab + Ibrutinib | Ibrutinib
All-Cause Mortality (participants affected / at risk) | 5/59 | 9/58
Serious Adverse Events (participants affected / at risk) | 38/59 | 31/58
Other Adverse Events (participants affected / at risk) | 59/59 | 57/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ublituximab + Ibrutinib (N=59) | Ibrutinib (N=58)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 1
Atrial fibrillation (Cardiac disorders) | 4 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Vitello-intestinal duct remnant (Congenital, familial and genetic disorders) | 1 | 0
Retinal tear (Eye disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 0
Fatigue (General disorders) | 0 | 1
Pneumonia (Infections and infestations) | 6 | 4
Sepsis (Infections and infestations) | 3 | 1
Cellulitis (Infections and infestations) | 2 | 0
Bacteraemia (Infections and infestations) | 1 | 1
Cellulitis staphylococcal (Infections and infestations) | 1 | 0
Meningitis aseptic (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 1
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0
Sinusitis bacterial (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Periorbital cellulitis (Infections and infestations) | 0 | 1
Periorbital infection (Infections and infestations) | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Incision site pain (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Gallbladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Bowens disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ublituximab + Ibrutinib (N=59) | Ibrutinib (N=58)
Increased tendency to bruise (Blood and lymphatic system disorders) | 2 | 3
Leukocytosis (Blood and lymphatic system disorders) | 2 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 12 | 4
Neutropenia (Blood and lymphatic system disorders) | 15 | 7
Anaemia (Blood and lymphatic system disorders) | 17 | 12
Atrial fibrillation (Cardiac disorders) | 5 | 4
Palpitations (Cardiac disorders) | 7 | 5
Dry eye (Eye disorders) | 5 | 2
Abdominal discomfort (Gastrointestinal disorders) | 2 | 3
Dysphagia (Gastrointestinal disorders) | 3 | 2
Oral pain (Gastrointestinal disorders) | 3 | 2
Haemorrhoids (Gastrointestinal disorders) | 4 | 1
Abdominal distension (Gastrointestinal disorders) | 5 | 1
Abdominal pain upper (Gastrointestinal disorders) | 5 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 4
Dry mouth (Gastrointestinal disorders) | 9 | 7
Abdominal pain (Gastrointestinal disorders) | 10 | 10
Dyspepsia (Gastrointestinal disorders) | 12 | 5
Stomatitis (Gastrointestinal disorders) | 12 | 7
Vomiting (Gastrointestinal disorders) | 13 | 4
Constipation (Gastrointestinal disorders) | 14 | 11
Nausea (Gastrointestinal disorders) | 24 | 19
Diarrhoea (Gastrointestinal disorders) | 34 | 26
Non-cardiac chest pain (General disorders) | 3 | 2
Influenza like illness (General disorders) | 4 | 4
Asthenia (General disorders) | 5 | 4
Pain (General disorders) | 5 | 3
Oedema peripheral (General disorders) | 11 | 16
Chills (General disorders) | 15 | 4
Pyrexia (General disorders) | 17 | 8
Fatigue (General disorders) | 23 | 22
Hypogammaglobulinaemia (Immune system disorders) | 9 | 3
Conjunctivitis (Infections and infestations) | 1 | 3
Eye infection (Infections and infestations) | 3 | 1
Fungal infection (Infections and infestations) | 3 | 0
Onychomycosis (Infections and infestations) | 3 | 1
Oral candidiasis (Infections and infestations) | 3 | 1
Paronychia (Infections and infestations) | 3 | 1
Skin infection (Infections and infestations) | 3 | 2
Ear infection (Infections and infestations) | 4 | 2
Influenza (Infections and infestations) | 4 | 1
Cellulitis (Infections and infestations) | 5 | 2
Herpes zoster (Infections and infestations) | 5 | 1
Bronchitis (Infections and infestations) | 6 | 2
Nasopharyngitis (Infections and infestations) | 6 | 5
Urinary tract infection (Infections and infestations) | 6 | 8
Pneumonia (Infections and infestations) | 11 | 5
Sinusitis (Infections and infestations) | 15 | 11
Upper respiratory tract infection (Infections and infestations) | 18 | 16
Procedural pain (Injury, poisoning and procedural complications) | 3 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 4 | 3
Skin abrasion (Injury, poisoning and procedural complications) | 4 | 2
Fall (Injury, poisoning and procedural complications) | 6 | 8
Contusion (Injury, poisoning and procedural complications) | 16 | 17
Infusion related reaction (Injury, poisoning and procedural complications) | 16 | 0
Blood bilirubin increased (Investigations) | 1 | 5
Alanine aminotransferase increased (Investigations) | 2 | 3
Aspartate aminotransferase increased (Investigations) | 2 | 3
Lymphocyte count increased (Investigations) | 3 | 2
Weight decreased (Investigations) | 4 | 3
Blood uric acid increased (Investigations) | 5 | 1
Blood creatinine increased (Investigations) | 7 | 2
Platelet count decreased (Investigations) | 8 | 8
Neutrophil count decreased (Investigations) | 9 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 3
Dehydration (Metabolism and nutrition disorders) | 3 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 8
Hyperuricaemia (Metabolism and nutrition disorders) | 5 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 7 | 6
Decreased appetite (Metabolism and nutrition disorders) | 10 | 7
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 5
Flank pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 14
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 13
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Neuropathy peripheral (Nervous system disorders) | 0 | 3
Paraesthesia (Nervous system disorders) | 5 | 2
Dysgeusia (Nervous system disorders) | 6 | 3
Dizziness (Nervous system disorders) | 15 | 15
Headache (Nervous system disorders) | 18 | 17
Confusional state (Psychiatric disorders) | 0 | 6
Depression (Psychiatric disorders) | 6 | 5
Anxiety (Psychiatric disorders) | 7 | 8
Insomnia (Psychiatric disorders) | 17 | 10
Urinary retention (Renal and urinary disorders) | 3 | 3
Haematuria (Renal and urinary disorders) | 4 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 9 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 25 | 18
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 3
Erythema (Skin and subcutaneous tissue disorders) | 2 | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 8
Onychoclasis (Skin and subcutaneous tissue disorders) | 4 | 3
Petechiae (Skin and subcutaneous tissue disorders) | 4 | 4
Ecchymosis (Skin and subcutaneous tissue disorders) | 5 | 5
Night sweats (Skin and subcutaneous tissue disorders) | 5 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 5
Skin lesion (Skin and subcutaneous tissue disorders) | 5 | 4
Rash (Skin and subcutaneous tissue disorders) | 8 | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 | 2
Flushing (Vascular disorders) | 3 | 1
Hot flush (Vascular disorders) | 4 | 3
Hypertension (Vascular disorders) | 8 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
TG Therapeutics has the right to review all proposed abstracts, manuscripts or presentations prior to submission for publication; however, the terms and conditions, including timing for review, of TG Therapeutics' agreements with its investigators may vary. Any single-site publications will be postponed until publication of data from the entire clinical trial (pooled from all sites). An investigator may not disclose TG Therapeutics confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-07-31): https://cdn.clinicaltrials.gov/large-docs/56/NCT02301156/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/56/NCT02301156/SAP_001.pdf